CLINICAL TRIAL: NCT06797089
Title: myTAP Oral Appliance Plus Mouth Shield to Reduce Periodontitis in Mouth-Breathers Who Snore
Brief Title: Does myTAP Oral Appliance Therapy Including a Mouth Shield Lessen Periodontitis in Mouth-Breathers Who Snore?
Acronym: OAplusPerio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2022-1450
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Snoring; Mouth Breathing; Daytime Sleepiness; Periodontitis
Keywords: Periodontitis; obstructive sleep apnea
MeSH Terms: conditions — Snoring; Mouth Breathing; Disorders of Excessive Somnolence; Periodontitis; Sleep Apnea, Obstructive | interventions — Weights and Measures

STUDY DESIGN:
Intervention Model Description: Oral Appliance plus mouth shield is applied to all subjects. Initially, all subjects will receive adjunctive scaling and root planing (SRP) on one side of the mouth (randomly assigned).
Masking Description: The periodontist performing the initial one-sided SRP does not know which side has been assigned to receive the therapy until the actual time of performance (blinding of investigator). The investigator is given an envelope with the side assignment at this time. Final assessment of periodontitis measures will be performed by a periodontist who will not be told which side of the mouth received the SRP therapy initially. Similarly, the investigator evaluating the oral bacteria samples will be blinded as to which side received SRP (blinding of outcomes assessors). The blinding pertains to the split-mouth design, not assignment of patients to treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- OA plus Mouth Shield (Experimental): Oral appliance therapy plus scaling and root planing on left or right of mouth
  Interventions: Device: Oral appliance therapy plus scaling and root planing on left or right of mouth

INTERVENTIONS:
Device: Oral appliance therapy plus scaling and root planing on left or right of mouth — This device opens the upper airway by bringing the mandible forward to improve breathing during sleep. The mouth shield minimizes mouth breathing to optimize salivary function. Scaling and root planing (deep cleaning of all teeth requiring it).
  Other Names: myTAP mandibular advancement device plus mouth shield

SUMMARY:
Mouth breathing, snoring and poor sleep can contribute to and worsen periodontitis (gum disease). The purpose of this study is to test whether the myTAP oral appliance with a mouth shield (OA+) can lessen periodontal symptoms in those with these conditions over a 12 week period. In addition to testing sleep respiration and quality, it will also evaluate periodontal pathogens and systemic stress in subjects treated with OA+. This split-mouth clinical trial will include adults with mild to moderate periodontist who snore and mouth breath. All will receive comprehensive periodontal care in addition to OA+ therapy.

DETAILED DESCRIPTION:
BACKGROUND & MOTIVATION

The keystone pathogen in chronic periodontitis, Porphyromonas gingivalis has been identified as a significant risk factor in the pathogenesis for developing Alzheimer's disease (AD) and was recently identified in the brains AD patients. Primary snoring, mouth breathing (MB) and obstructive sleep apnea (OSA) are also frequent findings in AD patients. MB impairs oral health, reduces quantity and quality of saliva, and increases dry mouth, risk of developing dental caries, gingival inflammation, bad breath and dry lips. This proposal aims to fill the information gap on the effects of oral appliance therapy on periodontitis by following up on participants in our previous randomized clinical trial.

INNOVATION

Periodontal disease affects about half of all US adults. Patients with periodontal inflammation, moderate to heavy bleeding of the gums with deep pockets demonstrate poor gum healing and persistent bacterial infection. Typically, patients are instructed to use over-the-counter oral rinse solutions twice a day to improve their periodontitis. OA used during sleep is expected to provide longer therapeutic exposure of saliva to teeth and gums in addition to optimizing upper airway stability, snoring and OSA attenuation, and MB inhibition.

DESCRIPTION

Two previous studies by the Sleep Research Program at Texas A&M University School of Dentistry have shown that with mandibular advancement oral appliance (OA) therapy, significant improvements in breathing during sleep and in cognition occur in those who have obstructive sleep apnea and snore. A third study suggests that improvements in the oral environment and in periodontal disease are possible with a combined therapy (OA+) that includes a mandibular advancement oral appliance with a mouth-shield (MS). The current study is intended to evaluate OA+ efficacy in attenuating mouth breathing and periodontal symptoms in those with these conditions over 12 weeks. In addition to testing sleep respiration and quality, it will also evaluate periodontal pathogens and systemic stress (assay using ELISA assay) in subjects treated with OA+. The clinical trial will include 27 adults with mild to moderate periodontist who snore and mouth breath. A randomized split-mouth design cohort design will be used to separate out the combined and independent effects of OA+ therapy and periodontal therapy. After an initial periodontal deep cleaning on one side of the mouth, all subjects will begin using an OA for 4 weeks. At 4 weeks, they will all begin using OA+ for the next 8 weeks. Changes from baseline to 4-, 8- and 12- weeks will be evaluated and compared on the periodontally treated and control sides. Their sleep respiration will be monitored using the NOX T3 sleep recorder for 1-night (pre-screening), and then 2 consecutive nights at baseline (T0) 4- 8- and 12 weeks Full periodontal evaluations will be performed at baseline, 4- 8- and 12 weeks. Plaque samples will be taken on both sides of the mouth at baseline and 12 weeks to evaluate periodontal and systemic pathogens. At the completion of the study, all subjects will receive a full mouth deep cleaning to optimize their periodontal health. As compensation, there will be no costs to participants for either the periodontal evaluation and treatment, or the OA+ therapy to improve their sleep. The myTAP OA, fabricated by AMI Inc. Dallas, TX will be the primary intervention. It is FDA cleared, low-cost, and is unique in that it includes a mouth-shield and is efficiently fitted chairside (no laboratory work or expenses involved). This dental care provided to participants at no cost to them would be approximately $750 at this dental school and up to $4500 in private practice.

Primary outcome variables: periodontal assessment, apnea hypopnea index, mouth breathing, respiration rate. Secondarily, Porphyromonas gingivalis and Aggregatibacter actinomycetemcomitans and cortisol will be assayed from plaque and saliva samples respectively. The projected timeline for the project is 12 months. Each subject will participate for 13-16 weeks.

The primary intervention, the myTAP oral appliance, and the sleep recorder , the NOX T3, are FDA cleared devices and have been in widespread use for many years.

ELIGIBILITY:
Inclusion Criteria:

1. Mouth breathing and snoring confirmed by home sleep test (NOX T3; ≥4 snores/hour) and complaints of excessive daytime sleepiness
2. Seeking treatment for periodontitis (stage 1 or 2 as confirmed by full periodontal examination at Visit 1 or 2)
3. Adults 18-85 years old
4. Stable medical condition (e.g., diabetes or hypertension properly managed)
5. At least 8 natural maxillary teeth to support the oral appliance
6. Mallampati score from I to III; Palatine tonsils - grade 0, 1, or 2
7. Central and mixed apnea index < 5 events/hour
8. Able to speak, read, and comprehend English fluently
9. At least 12 years of education
10. Ability to apply and remove home sleep recorder

    Willingness to...
11. Share PHI, medication list, current and past medical and dental information with research team members as needed
12. Follow all oral hygiene instructions and attend all appointments (periodontal and otherwise) as stipulated by the protocol
13. Allow the collection of plaque and waste materials from periodontal procedures and allow them to be evaluated for bacterial DNA (not human DNA)
14. Provide saliva samples (spit into tube)
15. Wear the oral appliance (OA) nightly as instructed for 12 weeks and with the mouth-shield (OA+) for the last 8 weeks
16. Complete brief surveys on sleep and related subjective experiences
17. Communicate with the clinical research coordinator regarding OA titration
18. Continue current medication and supplement use
19. Wait till the end of 12-week experimental period to complete periodontal therapy; this will include scaling, root planing of untreated side of dentition as well as redoing the treated side

Exclusion Criteria

1. Gingival probing depths > 5mm
2. Tooth mobility score greater than 2
3. Severe xerostomia
4. Severe medical illness such as symptomatic chronic obstructive pulmonary disease, renal failure, symptomatic coronary or cerebral vascular disease, cardiac dysrhythmia (i.e., atrial fibrillation); pacemaker; cardiopulmonary dysfunction (i.e., chronic heart failure),
5. Severe psychiatric and neurological disorders such as current substance abuse (including alcohol, nicotine); major depression and psychotic disorder; seizure disorder
6. Morbid obesity (Body Mass Index: BMI ≥35)
7. Active temporomandibular joint disorder (TMD) or jaw muscle pain; persistent history of TMD
8. Diagnosis of severe periodontitis
9. Morphological airway abnormalities (malformations of throat; e.g., a very small airway due to a condition such as severe micrognathia or Pierre Robin Syndrome)
10. Restrictions in jaw opening (difficult opening mouth widely) < 30 mm
11. Pre-existing difficulty swallowing; throat or neck related health issues;
12. Previous major surgery to throat and surrounding area such as UPPP (uvulopalatopharyngoplasty)
13. Intellectual disability that would prevent giving informed consent
14. Serious hormonal disease (endocrine dysfunction such as Addison's disease, Cushing's disease, hyperthyroidism); Diabetes and osteoporosis are OK)
15. Pregnant, breast feeding or intent to become pregnant during the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Periodontal conditions | Baseline to 3 months
  Periodontal condition staged (I-IV) according to The American Academy of Periodontology (AAP) 2018 Guidelines.
Mouth breathing | Baseline to 1, 2 and 3 months
  Presence of mouth breathing from NOX T3 sleep recording
Respiratory event index (REI) | Baseline to 1, 2 and 3 months
  Number of apneas and hypopneas per hour of recording from NOX T3 sleep recording
Respiration rate | Baseline to 1, 2 and 3 months
  Breaths per minute from NOX T3 sleep recording

SECONDARY OUTCOMES:
Periodontal and systemic bacteria from plaque samples | Baseline to 3 months
  Bacterial level in genome copies/milliliter in log10 values of 11 species
Mean oxygen desaturation, SaO2 | Baseline to 1, 2 and 3 months
  Mean percentage of oxygen saturation values obtained using pulse oximetry.
Salivary cortisol level | Baseline to 3 months
  Nanograms of cortisol per milliliter of saliva

CONTACTS AND LOCATIONS:
Overall Officials: Emet D Schneiderman, PhD, Principal Investigator — Texas A&M School of Dentistry
Locations (1):
- Texas A&M University College of Dentistry, Dallas, Texas, United States